CLINICAL TRIAL: NCT05456646
Title: The Change in Temporal Muscle Thickness and Its Relationship With Sarcopenia and Functional Outcomes in Stroke Patients.
Brief Title: The Change in Temporal Muscle Thickness in Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BITMS0722
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-01

CONDITIONS: Stroke; Sarcopenia
MeSH Terms: conditions — Stroke; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the relationship between sarcopenia and functional outcomes with temporal muscle mass change.

DETAILED DESCRIPTION:
It is well known that stroke increases the risk of developing sarcopenia . In addition, prestroke sarcopenia is associated with worse functional outcomes in patients with stroke. Temporal muscle thickness (TMT) has recently been proposed as a new marker of whole-body muscle mass and function. Measurement of temporal muscle mass by computed tomography (CT) and magnetic resonance imaging (MRI) has been studied in the literature in recent years. All stroke patients undergo cranial CT or MRI examinations at the time of admission. By evaluating the temporal muscle mass of these patients with these examinations, information about pre-stroke muscle mass and sarcopenia can be obtained. Ultrasonography (USG), on the other hand, may be a more accessible, less expensive, and safer option for assessing muscle mass in the follow-up of stroke patients. This study aims to evaluate the relationship between sarcopenia and functional outcomes with temporal muscle mass change by MRI/CT at admission and by USG in the chronic period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke
* Presence of cranial MRI/CT in hospital records

Exclusion Criteria:

* Medically unstable condition (presence or high risk of impaired consciousness, respiration, or circulation).
* Severe cognitive impairment
* Patients who require intensive care unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A tertiary health care facility
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Functional Ambulation Scale | Baseline
  This scale consists of six levels of function, ranging from 0 ( non-ambulatory ) to 5 (independently ambulatory).
Functional Ambulation Scale | 6. month
  This scale consists of six levels of function, ranging from 0 ( non-ambulatory ) to 5 (independently ambulatory).
The Functional Independence Measure (FIM) | Baseline
  FIM is a scale that assesses 18 activities, including self-care, sphincter control, transfer, movement, communication, and social awareness. Total scores range from 18 to 126 (dependent in all domains - independent in all domains).
The Functional Independence Measure (FIM) | 6.month
  FIM is a scale that assesses 18 activities, including self-care, sphincter control, transfer, movement, communication, and social awareness. Total scores range from 18 to 126 (dependent in all domains - independent in all domains).
Modified Rankin Scale (mRS) | Baseline
  It categorizes poststroke disability into six levels ranging from 0 to 5, with absence of symptoms rated as 0 and severe disability or bedriddenness rated as 5. An mRS score of 2 or less was defined as a good outcome, and an mRS score above 2 was defined as a poor outcome.
Modified Rankin Scale (mRS) | 6. month
  It categorizes poststroke disability into six levels ranging from 0 to 5, with absence of symptoms rated as 0 and severe disability or bedriddenness rated as 5. An mRS score of 2 or less was defined as a good outcome, and an mRS score above 2 was defined as a poor outcome.
Handgrip strength | Baseline
  With the JAMAR Hand Dynamometer, 3 measurements will be taken for both hands 60 seconds apart in the standard position and the highest reading will be recorded.
Handgrip strength | 6. month
  With the JAMAR Hand Dynamometer, 3 measurements will be taken for both hands 60 seconds apart in the standard position and the highest reading will be recorded.
Dual energy X-ray absorptiometry (DEXA) | Baseline
  DEXA can be used to determine lean body mass and total body fat. The appendicular skeletal mass index will be used in the evaluation of sarcopenia and in other analyzes.
Dual energy X-ray absorptiometry (DEXA) | 6.month
  DEXA can be used to determine lean body mass and total body fat. The appendicular skeletal mass index will be used in the evaluation of sarcopenia and in other analyzes.
Bioelectrical impedance analysis (BIA) | Baseline
  Body water mass, total body fat, and muscle mass can be determined with BIA.The appendicular skeletal mass index will be used in the evaluation of sarcopenia and in other analyzes.
Bioelectrical impedance analysis (BIA) | 6.month
  Body water mass, total body fat, and muscle mass can be determined with BIA.The appendicular skeletal mass index will be used in the evaluation of sarcopenia and in other analyzes.
Functional Oral Intake Scale | Baseline
  The scale is rated with values between 1 and 7. Level 1-3 refers to tube-dependent feeding, level 4-6 to full oral feeding with restrictions, and level 7 to oral feeding without restrictions.
Functional Oral Intake Scale | 6. month
  The scale is rated with values between 1 and 7. Level 1-3 refers to tube-dependent feeding, level 4-6 to full oral feeding with restrictions, and level 7 to oral feeding without restrictions.

CONTACTS AND LOCATIONS:
Overall Officials: Bugra Ince, MD, Principal Investigator — Izmir Bozyaka Education and Resarch Hospital
Locations (1):
- Izmir Bozyaka Research and Training Hostpital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
upon request

REFERENCES:
- [Background] Ryan AS, Ivey FM, Serra MC, Hartstein J, Hafer-Macko CE. Sarcopenia and Physical Function in Middle-Aged and Older Stroke Survivors. Arch Phys Med Rehabil. 2017 Mar;98(3):495-499. doi: 10.1016/j.apmr.2016.07.015. Epub 2016 Aug 13. PMID 27530769
- [Background] Nozoe M, Kanai M, Kubo H, Yamamoto M, Shimada S, Mase K. Prestroke sarcopenia and functional outcomes in elderly patients who have had an acute stroke: A prospective cohort study. Nutrition. 2019 Oct;66:44-47. doi: 10.1016/j.nut.2019.04.011. Epub 2019 Apr 25. PMID 31207438
- [Background] Nakanishi N, Okura K, Okamura M, Nawata K, Shinohara A, Tanaka K, Katayama S. Measuring and Monitoring Skeletal Muscle Mass after Stroke: A Review of Current Methods and Clinical Applications. J Stroke Cerebrovasc Dis. 2021 Jun;30(6):105736. doi: 10.1016/j.jstrokecerebrovasdis.2021.105736. Epub 2021 Mar 20. PMID 33756264